CLINICAL TRIAL: NCT00716261
Title: Using Bio-Feedback for Improving Stability in Walking and Everyday Activity
Brief Title: Bio-Feedback to Improving Stability in Elderly Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Laboratory for gait and neurodynamics, Tel Aviv Sourasky Medical center, Tel Aviv Sourasky Medical Center
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: 0204-08-TLV
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2008-07-16 (Estimated); Status verified 2008-07

CONDITIONS: Parkinson's Disease Patients
Keywords: Parkinson's disease; Audio feedback; postural control
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: McROB Hybrid node 3-axes accelerometers and 3-axes gyroscopes — Training with the Audio-feedback device for about 30 minutes, 3 times per week for 6 weeks
  Other Names: AUDIO-BIOFEEDBACK SYSTEM; DEIS, Università di Bologna; Bologna, Italy(Chiari et al., 2005)

SUMMARY:
Our hypothesis is that intensive training with positive biofeedback may enhance postural control and stability in Parkinson's disease patients and in elderly fallers.

DETAILED DESCRIPTION:
The aim of the study is to treat Parkinson's patients and elderly fallers. The intervention is intensive training with Biofeedback to try to correct stooped posture, and to improve stability in standing and in walking.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic PD for >2 yrs
* Between 50-90 Yrs
* On anti-Parkinsonian medication
* Hoehn & Yahr 2-3 in "ON"
* Free of serious co-morbidities
* Able to walk but reports difficulties in gait
* Can use assistive device

Exclusion Criteria:

* Significant orthopedic disturbances or pain
* Major depression (DSM IV)
* Dementia (MMSE<24)
* Clinically significant hearing problems
* Unstable medical condition (2 wks from meds change)
* Deep Brain Stimulation

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2008-01; Primary Completion 2009-09 (Estimated); Study Completion 2009-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Hausdorff, PhD, Principal Investigator — Laboratory for gait and neurodynamics, Tel-Aviv Sourasky Medical Center
Locations (1):
- Laboratory for gait and neurodynamics, Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel